CLINICAL TRIAL: NCT07327749
Title: Bisoprolol Monotherapy Versus Valsartan-Amlodipine for Hypertension Management in Adults Younger Than 60: Results of a Randomized Triple-Blind Clinical Trial
Brief Title: Comparing Bisoprolol and Valsartan-Amlodipine for Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SUMS.MED.REC.1402.206
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
Keywords: hypertension; bisoprolol; valsartan- amlodipine fix combination pill
MeSH Terms: conditions — Hypertension | interventions — Bisoprolol; Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bisoprolol (Active Comparator): Newly diagnosed hypertensives, proved by 24 hours holter monitoring, receiving tablet bisoprolol
  Interventions: Drug: Bisoprolol
- Valsartan- Amlodipine fix dose combination (Active Comparator): Newly diagnosed hypertensives, proved by 24 hours holter monitoring, receiving tablet valsartan-Amlodipine
  Interventions: Drug: valsartan and amlodipine

INTERVENTIONS:
Drug: Bisoprolol — Newly diagnosed hypertensives, proved by 24 hours holter monitoring, receiving tablet bisoprolol
  Other Names: concor
  Arms: bisoprolol
Drug: valsartan and amlodipine — Newly diagnosed hypertensives, proved by 24 hours holter monitoring, receiving tablet valsartan-amlodipine fix combination pill
  Other Names: valsartan-amlodipine fix combination pill
  Arms: Valsartan- Amlodipine fix dose combination

SUMMARY:
Randomized comparison of bisoprolol 2.5 mg monotherapy with fix combination drug valsartan 80 mg- amlodipine 5 mg

DETAILED DESCRIPTION:
In this randomized, triple-blind, two-arm clinical trial, 59 adults aged 18-60 years with newly diagnosed stage 1-2 hypertension were assigned to bisoprolol 2.5 mg once daily (n=30) or a valsartan 80 mg + amlodipine 5 mg single-pill combination (n=29) for two months. Blood pressure was assessed using 24-hour ambulatory monitoring at baseline and after treatment. Statistical analysis included paired t-tests, ANOVA, and nonparametric methods, with significance set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed stage 1 or stage 2 hypertension confirmed by 24-hour ambulatory blood pressure monitoring (ABPM).

Exclusion Criteria:

* Severe hypertension (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg)
* Contraindications to beta-blockers
* Contraindication to calcium channel blocker
* Contraindication to angiotensin receptor blockers
* Significant comorbidities requiring specific therapy such as diabetes or chronic heart failure, or current use of medications that could interact with the study drugs were excluded
* Pregnant or breastfeeding women
* Individuals with suspected secondary hypertension, and those unable to adhere to follow-up procedures

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
mean blood pressure | 2 months
  mean blood pressure derived from 24 hours holter monitoring
mean blood pressure nighttime | 2 months
  mean blood pressure at nighttime derived from 24 hours holter monitoring

SECONDARY OUTCOMES:
drug adverse effect | 2 months
  any drug adverse effect reported by patient

CONTACTS AND LOCATIONS:
Locations (1):
- professor Kojuri cardiology clinic, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
Data will be available with rational request